CLINICAL TRIAL: NCT00112203
Title: A Multicentre, Open-Label Extension Phase to Study the Long-Term Safety and Efficacy of Itopride HCl in Patients Suffering From Functional Dyspepsia
Brief Title: Long-Term Safety and Efficacy of Itopride Hydrochloride (HCl) in Patients Suffering From Functional Dyspepsia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Dr. M. Giguere, Axcan Pharma inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITOFD04-04
Record Dates: First submitted 2005-05-31; First posted 2005-06-01 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Dyspepsia
Keywords: Abdominal Symptom Relief; Fullness; Bloating; Indigestion; Functional dyspepsia
MeSH Terms: conditions — Dyspepsia | interventions — itopride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Itopride

SUMMARY:
Itopride is a compound already marketed in Japan and in some countries of Eastern Europe under the name of Ganaton. It is used to treat symptoms of functional dyspepsia. Patients suffering from this condition have difficulties digesting food. Patients feel full after eating; they have bloating and have stomach pain. The goal of this study is to see if itopride helps to relieve the symptoms of functional dyspepsia on a long-term basis.

DETAILED DESCRIPTION:
All patients who have completed study ITOFD04-03 will be offered to continue to be treated with itopride for a period of up to one year in duration. A target of 300 patients will be followed up for 6 months. Of these, a target of 100 patients will be kept on treatment for an additional 6 months.

Patients will need to come to the clinic for evaluations every 8 weeks during the trial. Evaluations done at these visits will include: lab tests, evaluation of the heartburn condition, and a questionnaire needed to be completed by the patient to see if the drug is helpful in relieving their symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have completed the 8 week double-blind study ITOFD04-03
* Female patients must not be pregnant (must have a negative serum pregnancy test)

Exclusion Criteria:

* Patients with any newly occurring medical condition which was an exclusion criterion at ITOFD04-03 study entry

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 466 (Actual)
Dates: Start 2004-11; Primary Completion 2006-07 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Long-term safety | every 2 months

SECONDARY OUTCOMES:
Long-term relief of symptoms | every 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Jan Tack, MD, Principal Investigator — University of Leuven

REFERENCES:
- [Derived] Broeders B, Tack J, Talley NJ. Itopride in functional dyspepsia: open-label, 1-year treatment follow-up of two multicenter, randomized, double-blind, placebo-controlled trials. Therap Adv Gastroenterol. 2025 Feb 20;18:17562848251321123. doi: 10.1177/17562848251321123. eCollection 2025. PMID 39989849